CLINICAL TRIAL: NCT02886520
Title: Multicentric Randomized Clinical Trial Comparing Polyvinylidene Fluoride and Polypropylene Transobturator Suburethral Tapes in the Treatment of Female Stress Urinary Incontinence.
Brief Title: Comparative Study of PDVF and Polypropylene Transobturator Suburethral Tapes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital de Granollers (Other); Hospital Quiron Sagrado Corazon (Other); Hospital de Mataró (Other); Hospital Riotinto (Unknown); Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitari de Bellvitge (Other); Hospital de Viladecans (Other); Hospital Santa Caterina (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(AMI)241-2015
Record Dates: First submitted 2016-08-27; First posted 2016-09-01 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Urinary Stress Incontinence
Keywords: Urinary incontinence; Materials; Surgery; Transobturator tape; Polyvinylidene fluoride; Polypropylene
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVDF transobturator tape (Active Comparator): Transobturator tension-free suburethral tape made of polyvinylidene fluoride.
  Interventions: Device: PVDF transobturator tape
- PP transobturator tape (Active Comparator): Transobturator tension-free suburethral tape made of polypropylene.
  Interventions: Device: Polypropylene transobturator tape

INTERVENTIONS:
Device: PVDF transobturator tape
  Other Names: Dynamesh-SIS
  Arms: PVDF transobturator tape
Device: Polypropylene transobturator tape
  Arms: PP transobturator tape

SUMMARY:
This study evaluates the effectiveness and complications of polyvinylidene fluoride (PVDF) and polypropylene (PP) transobturator suburethral tapes (TOTs) in the treatment of female stress urinary incontinence. Half of participants will be operated with PVDF-TOTs, while the other half will be operated with PP ones.

ELIGIBILITY:
Inclusion Criteria:

* Women with stress urinary incontinence.
* Women with stress-predominant mixed urinary incontinence.

Exclusion Criteria:

* Incapacity to understand the information or give their consent.
* Previous anti-incontinence surgery with slings.
* Low pressure urethra (MUCP < 20cmH2O).
* Neurogenic bladder.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness | One year
  Percentage of patients who are regarded as cured or improved one-year after surgery with both techniques based on the following criteria:
  * CURED: negative cough stress test and patient must be fully satisfied with the operation (no leaks, no voiding dysfunction, and no use of urinary protection); Patient Global Impresison of Improvement (PGI-I) scale must be "Very much better".
  * IMPROVED: cough stress test had to be negative and the patient moderately satisfied with the result of surgery due to an increase in urinary frequency and/or sporadic urgency episodes; PGI-I must be "Much better" or "A little better".

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to one year.
  Comparison of the intra- and postoperative complications between both procedures.

OTHER OUTCOMES:
Change in subjective questionnaires of incontinence severity | One year
  Change in the punctuation of the following questionnaires comparing before surgery and one year after operation:
  * International consultation on Incontinence Urinary Questionnaire-Short Form (ICIQ-SF).
  * Sandvik severity index.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital de Mataró, Barcelona
  - Hospital de Viladecans, Barcelona
  - Hospital General de Granollers, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Santa Caterina, Girona
  - Hospital General Riotinto, Huelva
  - Hospital Quiron Sagrado Corazon, Seville
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No